CLINICAL TRIAL: NCT00933114
Title: The Use of Functional Imaging to Quantify Tumor and Normal Tissue Physiology in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Functional Imaging of Tumor and Normal Tissue
Acronym: FITT
Status: Terminated | Type: Observational
Why Stopped: Funding ceased
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00014784
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Head and Neck Cancer
Keywords: DCE MRI; PET; Perfusion; Permeability; Cancer of the head and neck; Head, Neck neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Functional Imaging: Functional imaging with MRI and PET
  Interventions: Procedure: MRI and PET imaging

INTERVENTIONS:
Procedure: MRI and PET imaging — Dynamic Enhanced Magnetic Resonance Imaging (DEC-MRI) and positron emission tomography (PET) scan at baseline and after 1 week of radiation therapy

SUMMARY:
Dynamic contrast-enhanced (DCE) - magnetic resonance imaging (MRI), diffusion-weighted (DW)-MRI, and fludeoxyglucose - positron emission tomography - computed tomography (FDG-PET-CT) are three modalities that generate non-invasive, functional images of tumors and normal tissues based on physiologic properties including perfusion, vascular permeability and glucose metabolism. Demonstrating that these parameters are associated with clinical outcome, either efficacy or toxicity, could enhance the ability to select patients for different treatment strategies and improve the therapeutic ratio.

DETAILED DESCRIPTION:
Patients will undergo functional imaging studies, DCE-MRI pre-treatment (twice) and after 1 week of Radiation Therapy (RT) and PET scans - pre-treatment and after 1 week of RT. Parotid gland saliva production will also be measured at baseline and at 3, 6, and 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented squamous cell carcinoma of the head and neck (AJCC stages II-IV, M0)
* Eligible anatomic sites: Oral cavity, oropharynx, hypopharynx, supraglottic and glottic larynx, or nasopharynx
* Curative intent concurrent chemoradiation
* Age > 18 years
* Karnofsky Performance Status > 60
* Able to undergo MRI with contrast (gadolinium) and/or FDG PET scan

Exclusion Criteria:

* Diabetes other than diet controlled
* MRI Absolute Contraindications including:

  * Glomerular filtration rate < 60 ml/min
  * Weight < 350 lb or current device limitations
  * Metallic foreign bodies in the eye
  * Cardiac pacemakers
  * Clips in the central nervous system (ferromagnetic haemostatic)
  * Automatic internal cardiac defibrillators
  * Cochlear implants
  * Shrapnel in vital locations
* Pregnant (positive pregnancy test) or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to Radiation Oncology for radiotherapy of the NH cancer.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Permeability, perfusion, diffusion and glucose metabolism | At end of 1 week of radiation therapy

SECONDARY OUTCOMES:
Relationships between baseline and treatment induced changes in vascular permeability, perfusion, interstitial space, glucose metabolism, and saliva production to identify prognostic and predictive parameter(s) for treatment | 1 year of completing radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: David S Yoo, MD, PhD, Principal Investigator — Duke University Medical Center, Dept Radiation Oncology; David M Brizel, MD, Principal Investigator — Duke University Medical Center Dept Radiation Oncology
Locations (1):
- Duke University Medical Center, Department of Radiation Oncology, Durham, North Carolina, United States

REFERENCES:
- [Background] Brizel DM, Rosner GL, Prosnitz LR, Dewhirst MW. Patterns and variability of tumor oxygenation in human soft tissue sarcomas, cervical carcinomas, and lymph node metastases. Int J Radiat Oncol Biol Phys. 1995 Jul 15;32(4):1121-5. doi: 10.1016/0360-3016(95)00106-9. PMID 7607933
- [Background] Kirkpatrick JP, Cardenas-Navia LI, Dewhirst MW. Predicting the effect of temporal variations in PO2 on tumor radiosensitivity. Int J Radiat Oncol Biol Phys. 2004 Jul 1;59(3):822-33. doi: 10.1016/j.ijrobp.2004.02.015. PMID 15183486